CLINICAL TRIAL: NCT03092297
Title: Insufficient Cellular Oxygen in ICU Patients With Anaemia: the INOX ICU-2 Study
Brief Title: Insufficient Cellular Oxygen in ICU Patients With Anaemia
Acronym: INOX ICU-2
Status: Terminated | Type: Observational
Why Stopped: COVID-19 pandemic
Sponsor: Sanquin-LUMC J.J van Rood Center for Clinical Transfusion Research (Other)
Collaborators: Leiden University Medical Center (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Erasmus Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL59512.058.16
Record Dates: First submitted 2017-03-13; First posted 2017-03-27 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-12

CONDITIONS: Critical Care; Anemia; Erythrocyte Transfusion; Oxygen; Mitochondria
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be taken for measurement of: troponin, creatinine kinase, creatinine, hemoglobin, lactate, central venous oxygen saturation, arterial saturation, arterial oxygen tension, and venous oxygen tension. Remaining plasma will be frozen and stored for further evaulation
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ICU patients with anaemia: At admission to the ICU all patients, or their legal representatives, expected to stay at the ICU for longer than 24 hours will be asked to participate in the study and will be asked informed consent. ICU patients with anaemia in whom a central venous catheter is already in place and in whom a red cell transfusion is planned, will be included in the study.

SUMMARY:
The purpose of this study is whether the mitochondrial oxygenation tension (mitoPO2) is a feasible and reliable tool in ICU patients with anaemia undergoing red cell transfusion to ultimately personalize blood transfusion decisions in the ICU.

DETAILED DESCRIPTION:
Evidence is increasing that in some cases a Hb trigger of 7-8g/dl may be too low and te question arises whether an individualized red cell transfusion strategy may benefit critically ill patients. New studies have shown the potential of protoporphyrin IX-triple state lifetime technique to measure mitochondrial oxygenation tension (mitoPO2) in vivo, which possibly is an early indicator of oxygen disturbance in the cell and therefore a physiological trigger for red cell transfusion. The goals are: 1. Determining the feasibility of using mitoPO2 and the variability of mitoPO2 measurements in critically ill intensive care unit (ICU) patients before and after receiving a red cell transfusion 2. Describing the effects of red cell transfusion and the associated change in [Hb] on mitoPO2 and on other physiologic measures of tissue oxygenation and oxygen balance 3. Describing the association between mitoPO2 and vital organ functions. Included patients will undergo red cell transfusion as planned. However, red cell transfusion will be delayed by 2 hours. At multiple predefined moments data collection including blood samples and measurements of mitoPO2 will take place.

The results of this study cannot be immediately translated to clinical practice. Using these results, the investigators will design a phase 2 diagnostic study, most probably a randomized clinical trial that will yield applied knowledge with respect to personalizing red cell transfusion. Application will be in ICU patients with anaemia who might or might not profit from red cell transfusions. It will lead to a reduction of both over- and under- transfusion.

ELIGIBILITY:
Inclusion Criteria:

* adult patient admitted to the ICU
* Hb below 6.3 mmol/l (10 g/dl)
* central venous catheter in situ
* red cell transfusion planned

Exclusion Criteria:

* adults without a legal representative to ask for informed consent
* patients less than 18 years old
* pregnant or breast feeding women
* patients in need of emergency red cell transfusion e.g. bleeding
* not having a central venous catheter in situ
* porphyria and or known photodermatosis
* patients with an expected ICU stay <24 hours
* patients with hypersensitivity to the active substance or to the plaster material of ALA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted to the intensive care unit with a Hb below 6.3 mmol/l, with a central venous catheter in situ, who are planned to undergo a transfusion of red blood cells
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Variability of mitoPO2 | Variability of mitoPO2 will be assessed during 8 predefined moments (within a timeframe of 24 hours) in the study
  Variability of mitoPO2 before and after red cell transfusion. This will be compared to traditional parameters used to measure oxygenation and oxygen balance.

SECONDARY OUTCOMES:
Organ damage | Value of mitoPO2 in predicting (ischemic) organ damage will be assessed during 8 predefined moments (within a timeframe of 24 hours) in the study
  Value of mitoPO2 measurements for predicting (ischemic) organ damage
Microcirculation | Association of the mitoPO2 with the microcirculation will be assessed during 2 predefined moments (before transfusion and 24 hours after transfusion) in the study
  Association of mitoPO2 with the microcirculation
Length of stay | Length of stay will be assessed during the 3 months follow-up time
  Length of hospital-stay and ICu stay
Mortality | Mortality will be assessed during the 3 months follow-up time
  90-day mortality, hospital mortality and ICU mortality
Adverse events | Association of the mitoPO2 with adverse events will be assessed during 8 predefined moments (within a timeframe of 24 hours) in the study
  Adverse and serious adverse events of the mitoPO2 measurements

CONTACTS AND LOCATIONS:
Overall Officials: Johanna G van der Bom, PhD, MD, Study Chair — Leiden University Medical Center and Sanquin Research Leiden; M S Arbous, PhD, MD, Study Chair — Leiden University Medical Center; M Baysan, MD, Principal Investigator — Leiden University Medical Center and Sanquin Research Leiden
Locations (2):
- Netherlands (2):
  - Amsterdam Medical Center, Amsterdam, Amsterdam-Zuidoost, Noord-Holland
  - Leiden University Medical Center, Leiden, South Holland

IPD SHARING:
Plan to Share IPD: Undecided
to be decided

REFERENCES:
- [Derived] Baysan M, Hilderink B, van Manen L, Caram-Deelder C, Mik EG, Juffermans NP, van der Bom JG, Arbous MS. Mitochondrial oxygen tension in critically ill patients receiving red blood cell transfusions: a multicenter observational cohort study. Intensive Care Med Exp. 2024 Jul 8;12(1):61. doi: 10.1186/s40635-024-00646-3. PMID 38976096
- [Derived] Baysan M, Arbous MS, Mik EG, Juffermans NP, van der Bom JG. Study protocol and pilot results of an observational cohort study evaluating effect of red blood cell transfusion on oxygenation and mitochondrial oxygen tension in critically ill patients with anaemia: the INsufficient Oxygenation in the Intensive Care Unit (INOX ICU-2) study. BMJ Open. 2020 May 17;10(5):e036351. doi: 10.1136/bmjopen-2019-036351. PMID 32423938

DOCUMENTS (1):
  • Study Protocol (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/97/NCT03092297/Prot_001.pdf